CLINICAL TRIAL: NCT07023536
Title: Evaluation of the Effectiveness of a Cardiac Telerehabilitation Program in Chronic Heart Failure
Brief Title: Effectiveness of a Cardiac Telerehabilitation Program in Chronic Heart Failure
Acronym: TELEREHAB-HF
Status: Not yet recruiting | Type: Observational
Sponsor: University of Salerno (Other)
Collaborators: Azienda Ospedaliera OO.RR. S. Giovanni di Dio e Ruggi D'Aragona (Other)
Responsible Party: Principal Investigator, Alessia Bramanti, Associate Professor, University of Salerno
Other Study IDs: UNISA-TELEREHABHF-2025
Record Dates: First submitted 2025-06-08; First posted 2025-06-17 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure
Keywords: Chronic Heart Failure; Cardiac Rehabilitation; Tele-rehabilitation; Telemedicine; Exercise Training; Remote Monitoring; mHealth; Wearable Sensors; Home-based Rehabilitation; Digital Health
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The study will collect and retain the following biospecimens from participants for clinical and research purposes:
  Types of Samples Retained:
  Blood Samples
  * Plasma and serum - for analysis of biochemical markers related to chronic heart failure (e.g., B-type Natriuretic Peptide [BNP], N-terminal pro-B-type Natriuretic Peptide [NT-proBNP], creatinine, electrolytes, glucose, and lipid profile)
  * Urine Samples - To assess kidney function and electrolyte balance. All biospecimens will be pseudo-anonymized and stored securely following ethical guidelines (EU GDPR 2016/679) and institutional biobank policies. Participants will provide specific informed consent for sample retention and potential future research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- TELEREHABILITATION-YES (Intervention Group): Participants will receive a structured 8-week cardiac rehabilitation program conducted entirely at home through a certified telehealth platform (Khymeia VRRS system). The intervention includes real-time supervision by a physiotherapist via videoconferencing, and the use of wearable medical devices for continuous monitoring of vital signs (ECG, heart rate, SpO₂, blood pressure) and motion tracking. Each session includes warm-up, endurance training, and cooldown exercises, with intensity personalized based on baseline cardiopulmonary testing. The platform provides automated data recording, safety alerts, and performance feedback to ensure high-quality remote care. Patients are trained in-person before starting home-based sessions to ensure proper use of the system and adherence to the protocol.
  Interventions: Behavioral: TELEREHABILITATION-YES
- TELEREHABILITATION-NO (Control Group): Participants in this group will undergo a standard 8-week cardiac rehabilitation program delivered in person at the outpatient facility under direct supervision of a physiotherapist. This group receives face-to-face rehabilitation consisting of individualized exercise sessions performed at the hospital's cardiac rehabilitation unit. Each session includes warm-up, endurance training on a stationary bike, and cooldown, following international guidelines for heart failure patients. Vital signs (heart rate, blood pressure, oxygen saturation) are manually measured and recorded by the physiotherapist, who also administers fatigue and dyspnea scales (Borg and Rate of Perceived Exertion - RPE) throughout the program. No wearable technology is used in this group; monitoring is performed through direct clinical observation and documentation in the medical record.
  Interventions: Behavioral: TELEREHABILITATION-NO

INTERVENTIONS:
Behavioral: TELEREHABILITATION-YES — This intervention consists of a structured 8-week cardiac rehabilitation program performed at the patient's home using a certified telemedicine platform. Sessions are delivered in synchronous mode with real-time supervision by a physiotherapist through secure video conferencing. Each session includes warm-up, endurance training, and cooldown exercises, with personalized intensity based on cardiopulmonary exercise testing. Patients are equipped with wearable medical devices for continuous monitoring of vital signs (ECG, heart rate, blood pressure, oxygen saturation) and motion sensors to assess exercise execution and adherence. All data are transmitted securely and stored automatically in the system's database. In addition to the exercise protocol, participants undergo baseline and follow-up assessments including blood biomarkers, echocardiography, cardiopulmonary exercise testing, and quality-of-life questionnaires.
  Groups: TELEREHABILITATION-YES (Intervention Group)
Behavioral: TELEREHABILITATION-NO — This intervention involves a traditional 8-week cardiac rehabilitation program carried out at a hospital-based outpatient facility. Patients attend sessions in person under the direct supervision of a physiotherapist. Each session includes warm-up, endurance training using a stationary bike, and cooldown. Vital signs (e.g., heart rate, blood pressure, oxygen saturation) are monitored manually by the physiotherapist, and exercise tolerance is assessed using standardized clinical scales (e.g., Borg and RPE). In addition to the exercise protocol, participants undergo baseline and follow-up assessments including blood biomarkers, echocardiography, cardiopulmonary exercise testing, and validated quality-of-life questionnaires. This group serves as the control for evaluating the effectiveness of the home-based telerehabilitation model.
  Groups: TELEREHABILITATION-NO (Control Group)

SUMMARY:
The goal of this observational study is to evaluate whether a home-based cardiac tele-rehabilitation program can improve functional capacity in adults (18 years and older) with chronic heart failure. The main questions it aims to answer are:

Does tele-rehabilitation improve peak oxygen uptake (VO₂ max) compared to standard in-hospital rehabilitation? Does it improve cardiac function, exercise tolerance, biochemical markers, and quality of life? Are functional gains maintained at 24 weeks? Researchers will compare patients who opt for tele-rehabilitation using wearable devices and a remote monitoring platform with those undergoing standard in-person rehabilitation. Participants will follow an 8-week individualized training program and undergo assessments at baseline, 4, 8, 16, and 24 weeks.

DETAILED DESCRIPTION:
This prospective, single-center, non-pharmacological observational study aims to evaluate the effectiveness and feasibility of a structured, home-based cardiac telerehabilitation program in adults with chronic heart failure (CHF). The primary objective is to determine whether a telemedicine-based model can improve patients' functional capacity, as measured by maximal oxygen uptake (VO₂max), when compared to conventional in-hospital cardiac rehabilitation.

Participants will voluntarily enroll in either the telerehabilitation group or the standard rehabilitation group. Both groups follow the same 8-week aerobic exercise protocol, based on current international guidelines for heart failure management. The program includes warm-up, interval and endurance training, and cooldown, with exercise intensity personalized using cardiopulmonary exercise testing (CPET).

The telerehabilitation group will perform all sessions at home using a certified telehealth platform (Khymeia Virtual Reality Rehabilitation System - VRRS), which enables real-time supervision via secure videoconferencing. Participants are equipped with wearable medical-grade sensors for continuous monitoring of electrocardiogram (ECG), heart rate, blood pressure, and peripheral capillary oxygen saturation (SpO₂). The system offers automated data recording, performance feedback, and safety alerts, ensuring standardized care delivery and real-time clinical oversight. Before home-based training begins, participants receive structured in-person training to ensure safe and effective use of the digital tools.

Clinical and functional data are collected at baseline and follow-up visits at 4, 8, 16, and 24 weeks. The study also investigates patient adherence, safety, and the usability of digital rehabilitation tools. No investigational drugs or invasive procedures are involved. The findings will inform future implementation of scalable digital rehabilitation models in heart failure management and contribute to health system innovation in chronic disease care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of chronic heart failure for at least 6 months, with stable optimal medical therapy for at least 1 month
* New York Heart Association (NYHA) functional class I, II, or III
* Hospitalization or outpatient visit requiring intravenous therapy (diuretics, vasodilators, or inotropes) within the past 12 months
* Ability to provide informed consent or presence of a legal representative
* Digital literacy of the patient and/or caregiver

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* NYHA class IV heart failure
* Severe renal insufficiency (eGFR <30 ml/min/1.73 m²) or on dialysis
* Other serious illnesses significantly limiting life expectancy (e.g., end-stage cancer, advanced pulmonary disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: dults aged 18 years or older with a diagnosis of chronic heart failure, including heart failure with reduced ejection fraction (HFrEF), mildly reduced ejection fraction (HFmrEF), or preserved ejection fraction (HFpEF), and classified as NYHA functional class I to III, referred for cardiac rehabilitation at a tertiary care center. Participants must be clinically stable, receiving optimal medical therapy, and able to participate in either an in-person or home-based telerehabilitation program. Digital literacy, either of the patient or a caregiver, is required for inclusion in the telerehabilitation group. Both sexes are included. Patients with severe comorbidities that significantly limit life expectancy or with NYHA class IV heart failure are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 205 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in VO₂max from baseline to 8 weeks | Baseline (T=0) and end of intervention (T=2, 8 weeks)
  The primary outcome is the change in maximal oxygen consumption (VO₂max) from baseline to 8 weeks in patients with chronic heart failure undergoing a cardiac telerehabilitation program compared to a traditional in-person rehabilitation program. VO₂max is assessed via cardiopulmonary exercise testing (CPET). The intervention aims to achieve a clinically meaningful increase of approximately 20% in VO₂max. VO₂max is a key marker of functional capacity and cardiovascular health, and its improvement is associated with better prognosis, reduced hospitalizations, and enhanced quality of life.

SECONDARY OUTCOMES:
VO₂max at 24-week follow-up | follow-up (T=4, 24 weeks)
  This outcome assesses VO₂max measured at 24 weeks following the end of the intervention period, in order to evaluate the evolution of functional capacity over time. VO₂max is assessed using cardiopulmonary exercise testing (CPET) at baseline, 8 weeks, and 24 weeks. The analysis will examine whether any changes observed after the intervention are sustained, reversed, or further modified at follow-up.
Change in functional capacity assessed by 6-minute walk test (6MWT) | Baseline (T=0), 4 weeks (T=1), 8 weeks (T=2), 16 weeks (T=3), 24 weeks (T=4)
  Functional capacity will be measured using the 6-minute walk test (6MWT), a validated submaximal exercise test in heart failure patients. The distance walked will be recorded at baseline, after the 8-week intervention, and at 24-week follow-up. Improvements in distance will reflect better exercise tolerance, which is a relevant indicator of clinical status and therapeutic efficacy.
Change in Quality of Life | Baseline (T=0), 4 weeks (T=1), 8 weeks (T=2), 16 weeks (T=3), 24 weeks (T=4)
  Quality of life (QoL) will be measured using the Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall Summary Score, a validated instrument specifically designed to assess symptom burden, functional status, social limitations, and quality of life in patients with chronic heart failure (CHF). The score ranges from 0 to 100, where higher scores indicate better health status and quality of life.
Change in Quality of Life | Baseline (T=0), 4 weeks (T=1), 8 weeks (T=2), 16 weeks (T=3), 24 weeks (T=4)
  The Short Form Health Survey - 36 items (SF-36) evaluates general health status across multiple domains, including physical functioning, role limitations, pain, general health, vitality, social functioning, emotional well-being, and mental health. The total score ranges from 0 to 100, with higher scores indicating better health status and quality of life.
Change in Biochemical Parameters | Baseline (T=0), 8 weeks (T=2), 16 weeks (T=3), 24 weeks (T=4)
  Biochemical Parameters: Change in B-type Natriuretic Peptide (BNP) Levels (picograms per milliliter)
Change in Biochemical Parameters | Baseline (T=0), 8 weeks (T=2), 16 weeks (T=3), 24 weeks (T=4)
  Biochemical Parameters: Change in N-terminal pro-BNP (NT-proBNP) Levels (picograms per milliliter)
Change in Biochemical Parameters | Baseline (T=0), 8 weeks (T=2), 16 weeks (T=3), 24 weeks (T=4)
  Biochemical Parameters: Change in Serum Creatinine (milligrams per deciliter)
Change in Biochemical Parameters | Baseline (T=0), 8 weeks (T=2), 16 weeks (T=3), 24 weeks (T=4)
  Biochemical Parameters: Change in Estimated Glomerular Filtration Rate (eGFR) (milliliters per minute per 1.73 square meters)
Change in Biochemical Parameters | Baseline (T=0), 8 weeks (T=2), 16 weeks (T=3), 24 weeks (T=4)
  Biochemical Parameters: Change in Serum Sodium Levels (millimoles per liter)
Change in Biochemical Parameters | Baseline (T=0), 8 weeks (T=2), 16 weeks (T=3), 24 weeks (T=4)
  Biochemical Parameters: Change in Serum Potassium Levels (millimoles per liter)
Change in Biochemical Parameters | Baseline (T=0), 8 weeks (T=2), 16 weeks (T=3), 24 weeks (T=4)
  Biochemical Parameters: Change in Serum Chloride Levels (millimoles per liter)
Change in Functional ECG-Derived Parameters | Baseline (T=0), 8 weeks (T=2), 16 weeks (T=3), 24 weeks (T=4)
  ECG-Derived Parameters: Change in Heart Rate Variability (HRV) (milliseconds)
Change in Functional ECG-Derived Parameters | Baseline (T=0), 8 weeks (T=2), 16 weeks (T=3), 24 weeks (T=4)
  ECG-Derived Parameters: Change in Respiratory Rate (breaths per minute)
Change in Functional Echocardiographic derived Parameters | Baseline (T=0), 8 weeks (T=2), 16 weeks (T=3), 24 weeks (T=4)
  Echocardiographic Parameters: Change in Left Ventricular Ejection Fraction (LVEF) (percent)
Change in Functional Echocardiographic derived Parameters | Baseline (T=0), 8 weeks (T=2), 16 weeks (T=3), 24 weeks (T=4)
  Echocardiographic Parameters: Change in Diastolic Function - E/A Ratio (unitless)
Change in Functional Echocardiographic derived Parameters | Baseline (T=0), 8 weeks (T=2), 16 weeks (T=3), 24 weeks (T=4)
  Echocardiographic Parameters: Change in Left Ventricular End-Diastolic Volume (milliliters)
Change in Functional Echocardiographic derived Parameters | Baseline (T=0), 8 weeks (T=2), 16 weeks (T=3), 24 weeks (T=4)
  Echocardiographic Parameters: Change in Left Ventricular End-Systolic Volume (milliliters)
Change in cognitive function assessed by Mini-Mental State Examination (MMSE) | Baseline (T=0), 4 weeks (T=1), 8 weeks (T=2), 16 weeks (T=3), 24 weeks (T=4)
  Cognitive function will be assessed using the Mini-Mental State Examination (MMSE), a widely used screening tool for cognitive impairment. The MMSE evaluates orientation, attention, memory, language, and visuospatial skills. The total score ranges from 0 to 30, with higher scores indicating better cognitive function. Scores will be collected to monitor changes in cognitive status over time in patients participating in the cardiac rehabilitation program.
Change in physical performance assessed by Short Physical Performance Battery (SPPB) | Baseline (T=0), 4 weeks (T=1), 8 weeks (T=2), 16 weeks (T=3), 24 weeks (T=4)
  Change in physical performance will be assessed using the Short Physical Performance Battery (SPPB), which includes tests of balance, gait speed, and chair stands. The SPPB provides a composite score ranging from 0 to 12, with higher scores indicating better lower extremity function and physical performance.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heidenreich PA, Bozkurt B, Aguilar D, Allen LA, Byun JJ, Colvin MM, Deswal A, Drazner MH, Dunlay SM, Evers LR, Fang JC, Fedson SE, Fonarow GC, Hayek SS, Hernandez AF, Khazanie P, Kittleson MM, Lee CS, Link MS, Milano CA, Nnacheta LC, Sandhu AT, Stevenson LW, Vardeny O, Vest AR, Yancy CW; ACC/AHA Joint Committee Members. 2022 AHA/ACC/HFSA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2022 May 3;145(18):e895-e1032. doi: 10.1161/CIR.0000000000001063. Epub 2022 Apr 1. PMID 35363499
- [Background] Visseren FLJ, Mach F, Smulders YM, Carballo D, Koskinas KC, Back M, Benetos A, Biffi A, Boavida JM, Capodanno D, Cosyns B, Crawford C, Davos CH, Desormais I, Di Angelantonio E, Franco OH, Halvorsen S, Hobbs FDR, Hollander M, Jankowska EA, Michal M, Sacco S, Sattar N, Tokgozoglu L, Tonstad S, Tsioufis KP, van Dis I, van Gelder IC, Wanner C, Williams B; ESC National Cardiac Societies; ESC Scientific Document Group. 2021 ESC Guidelines on cardiovascular disease prevention in clinical practice. Eur Heart J. 2021 Sep 7;42(34):3227-3337. doi: 10.1093/eurheartj/ehab484. No abstract available. PMID 34458905
- [Background] Sui X, Gutekunst WR. Cascade Alternating Metathesis Cyclopolymerization of Diynes and Dihydrofuran. ACS Macro Lett. 2022 May 17;11(5):630-635. doi: 10.1021/acsmacrolett.2c00140. Epub 2022 Apr 18. PMID 35570817
- [Background] Sullivan DJ Jr. A Single Human Cerebral Malaria Histopathologic Study Can Be Worth a Thousand Experiments. mBio. 2015 Nov 17;6(6):e01818-15. doi: 10.1128/mBio.01818-15. PMID 26578683
- [Background] Taylor RS, Dalal HM, Zwisler AD. Cardiac rehabilitation for heart failure: 'Cinderella' or evidence-based pillar of care? Eur Heart J. 2023 May 1;44(17):1511-1518. doi: 10.1093/eurheartj/ehad118. PMID 36905176
- [Background] Flynn KE, Pina IL, Whellan DJ, Lin L, Blumenthal JA, Ellis SJ, Fine LJ, Howlett JG, Keteyian SJ, Kitzman DW, Kraus WE, Miller NH, Schulman KA, Spertus JA, O'Connor CM, Weinfurt KP; HF-ACTION Investigators. Effects of exercise training on health status in patients with chronic heart failure: HF-ACTION randomized controlled trial. JAMA. 2009 Apr 8;301(14):1451-9. doi: 10.1001/jama.2009.457. PMID 19351942
- [Background] Taylor RS, Walker S, Smart NA, Piepoli MF, Warren FC, Ciani O, Whellan D, O'Connor C, Keteyian SJ, Coats A, Davos CH, Dalal HM, Dracup K, Evangelista LS, Jolly K, Myers J, Nilsson BB, Passino C, Witham MD, Yeh GY; ExTraMATCH II Collaboration. Impact of Exercise Rehabilitation on Exercise Capacity and Quality-of-Life in Heart Failure: Individual Participant Meta-Analysis. J Am Coll Cardiol. 2019 Apr 2;73(12):1430-1443. doi: 10.1016/j.jacc.2018.12.072. PMID 30922474
- [Background] Taylor RS, Long L, Mordi IR, Madsen MT, Davies EJ, Dalal H, Rees K, Singh SJ, Gluud C, Zwisler AD. Exercise-Based Rehabilitation for Heart Failure: Cochrane Systematic Review, Meta-Analysis, and Trial Sequential Analysis. JACC Heart Fail. 2019 Aug;7(8):691-705. doi: 10.1016/j.jchf.2019.04.023. Epub 2019 Jul 10. PMID 31302050
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Background] Isernia S, Pagliari C, Morici N, Toccafondi A, Banfi PI, Rossetto F, Borgnis F, Tavanelli M, Brambilla L, Baglio F; CPTM Group. Telerehabilitation Approaches for People with Chronic Heart Failure: A Systematic Review and Meta-Analysis. J Clin Med. 2022 Dec 21;12(1):64. doi: 10.3390/jcm12010064. PMID 36614865
- [Background] Burns RB, Crislip D, Daviou P, Temkin A, Vesmarovich S, Anshutz J, Furbish C, Jones ML. Using telerehabilitation to support assistive technology. Assist Technol. 1998;10(2):126-33. doi: 10.1080/10400435.1998.10131970. PMID 10339280
- [Background] Jansen-Kosterink S, In 't Veld RH, Hermens H, Vollenbroek-Hutten M. A Telemedicine Service as Partial Replacement of Face-to-Face Physical Rehabilitation: The Relevance of Use. Telemed J E Health. 2015 Oct;21(10):808-13. doi: 10.1089/tmj.2014.0173. Epub 2015 Jun 4. PMID 26431260
- [Derived] Garofano M, Vecchione C, Calabrese M, Rusciano MR, Visco V, Granata G, Carrizzo A, Galasso G, Bramanti P, Corallo F, Pepe L, Budaci L, Ciccarelli M, Bramanti A. Evaluation of the Effectiveness of a Cardiac Telerehabilitation Program in Chronic Heart Failure: Design and Rationale of the TELEREHAB-HF Study. Healthcare (Basel). 2025 Aug 21;13(16):2074. doi: 10.3390/healthcare13162074. PMID 40868691